CLINICAL TRIAL: NCT03994081
Title: Mechanism of Action for Transcranial Alternating Current (tACS) Stimulation for the Treatment of Major Depressive Disorder (MDD)
Brief Title: Mechanism of Action of tACS for the Treatment of MDD
Acronym: GLADIATOR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Foundation of Hope, North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20-1822
Record Dates: First submitted 2019-06-10; First posted 2019-06-21 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Disorder; MDD
Keywords: tACS; Major Depressive Disorder; MDD; mood symptoms; sham
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Using sham stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- alpha Transcranial alternating current stimulation (tACS). (Experimental): 10 Hz tACS with a zero-to-peak amplitude of 1 mA for 40 minutes.
  Interventions: Device: tACS
- Sham stimulation (Sham Comparator): 20 seconds of ramp-up, 40 seconds of 10 Hz tACS with zero-to-peak amplitude of 1 mA, and 20 seconds of ramp-down for a total of 80 seconds of stimulation.
  Interventions: Device: Sham tACS

INTERVENTIONS:
Device: tACS — XCSITE100
  Arms: alpha Transcranial alternating current stimulation (tACS).
Device: Sham tACS — XCSITE100
  Arms: Sham stimulation

SUMMARY:
The purpose of this research study is to use a specific type of non-invasive brain stimulation known as transcranial alternating current stimulation (tACS) to determine its effects on brain activity (measured with EEG) and mood in patients with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
The device used for non-invasive brain stimulation is investigational and has not been approved by the FDA, though it has been designated as a nonsignificant risk (NSR) device study by the FDA. Half of the participants will receive tACS and half will receive sham stimulation, an inactive control procedure for comparison use only. Participation in this study includes up to eight appointments, each one lasting from 30 minutes to four hours over the course of 3 weeks. The first two appointments will be remote interviews to determine eligibility. If the subjects qualify, the next five appointments will be scheduled as consecutive stimulation sessions in the Carolina Center for Neurostimulation at the Vilcom office. The follow-up appointment will be in our center two weeks after the completion of the stimulation sessions. We estimate the total time needed to complete study participation to be about 17 hours.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years
* DSM-IV diagnosis of MDD; unipolar, non-psychotic
* Hamilton Rating Depression Rating Scale (HRDS-17) score >8
* Low suicide risk as determined by a score of <3 on the Suicide Item on the HDRS-17 and based on additional information from the C-SSRS (no intent)
* Capacity to understand all relevant risks and potential benefits of the study (informed consent)

Exclusion Criteria:

* DSM-V diagnosis of moderate or severe alcohol use disorder (AUD) within the last 12 months.
* DSM-V diagnosis of moderate to severe substance use disorder (excluding tobacco) within the last 12 months.
* Current axis I mood, or psychotic disorder other than major depressive disorder
* Lifetime comorbid psychiatric bipolar or psychotic disorder
* Eating disorder (current or within the past 6 months)
* Obsessive-compulsive disorder (lifetime)
* Post-traumatic stress disorder (PTSD, current or within the last 6 months)
* Change of ADHD medication within the last 4 weeks.
* Change of benzodiazepines or anti-epileptic medication within the last 4 weeks
* Antidepressant drugs taken for less than 4 weeks (i.e., recently initiated)
* Neurological disorders, including but not limited to history of seizures (except childhood febrile seizures and ECT-induced seizures), dementia, history of stroke, Parkinson's disease, multiple sclerosis, cerebral aneurysm.
* Medical or neurological illness (unstable cardiac disease, AIDS, malignancy, liver or renal impairment) or treatment for a medical disorder that could interfere with study participation; comorbid neurological condition (i.e. seizure disorder, brain tumor)
* History of traumatic brain injury that required subsequent cognitive rehabilitation, or cause cognitive sequelae.
* Prior brain surgery and/or any brain devices/implants, including cochlear implants and aneurysm clips
* Current pregnancy or lactation. If the ability to become pregnant exists, unwillingness to use appropriate birth control measures during study participation
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study
* Non-English speakers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rubinow, MD, Principal Investigator — University of North Carolina at Chapel Hill - Department of Psychiatry
Locations (1):
- UNC at Vilcom Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be available starting from 9 to 36 months following publication.
Access Criteria: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alpha Transcranial Alternating Current Stimulation (tACS) | Sham Stimulation
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpha Transcranial Alternating Current Stimulation (tACS) | Sham Stimulation | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 6 | 12
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in the Amplitude of Left Frontal Alpha Oscillations Measured Durin Resting-state EEG Recordings From Baseline to Day 5 of Stimulation.
Description: Fourier transform is applied to 2 second epochs of resting-state EEG data and averaged across epochs. The amplitude of alpha oscillations is calculated and averaged across left frontal electrodes. The difference between the baseline recording on the first day of stimulation is compared to the recording on the fifth day of the intervention prior to stimulation.
Time Frame: Baseline, Day 5
Population: Day 5 - Day 1
Measure: Mean (Standard Deviation); unit: microvolts^2/Hz
Arm/Group | Alpha Transcranial Alternating Current Stimulation (tACS) | Sham Stimulation
Number analyzed (Participants) | 10 | 10
microvolts^2/Hz | 0.042 (0.221) | 0.169 (0.338)
Statistical Analysis 1: Comparison: Alpha Transcranial Alternating Current Stimulation (tACS) vs Sham Stimulation; Test type: Superiority; p = 0.332, t-test, 2 sided

2. Primary Outcome: Change in the Amplitude of Left Frontal Alpha Oscillations Measured During Resting-state EEG Recordings From Baseline to Two-week Follow-up of Stimulation.
Description: Fourier transform is applied to 2 second epochs of resting-state EEG data and averaged across epochs. The amplitude of alpha oscillations is calculated and averaged across left frontal electrodes. The difference between the baseline recording on the first day of stimulation is compared to the recording on the two-week follow-up after intervention.
Time Frame: Baseline, two-week follow-up visit
Population: Data for 1 participant unavailable due to missed visit.
Measure: Mean (Standard Deviation); unit: microvolts^2/Hz
Arm/Group | Alpha Transcranial Alternating Current Stimulation (tACS) | Sham Stimulation
Number analyzed (Participants) | 9 | 10
microvolts^2/Hz | -0.016 (0.199) | 0.012 (0.243)
Statistical Analysis 1: Comparison: Alpha Transcranial Alternating Current Stimulation (tACS) vs Sham Stimulation; Test type: Superiority; p = 0.790, t-test, 2 sided

3. Secondary Outcome: Correlation Between Changes in the Amplitude of Left Frontal Alpha Oscillations From Baseline to Day 5 of Intervention and Changes in Symptoms of Depression.
Description: Correlation Coefficient (r) will be used to determine if there is a relationship between the change in Hamilton Depression Rating Scale (HDRS) scores from baseline to Day 5 and the two-week follow up and change in the amplitude of left frontal alpha oscillations before stimulation at baseline and Day 5 of stimulation. The HDRS is a clinician-rated measure of depression severity where higher scores indicate greater depression severity. To calculate the amplitude of left frontal alpha oscillations, Fourier transform is applied to 2 second epochs of resting-state EEG data and averaged across epochs. The amplitude of alpha oscillations is calculated and averaged across left frontal electrodes.
Time Frame: Baseline, Day 5
Measure: Number; unit: Pearson Correlation Coefficient
Arm/Group | Alpha Transcranial Alternating Current Stimulation (tACS) | Sham Stimulation
Number analyzed (Participants) | 10 | 10
Pearson Correlation Coefficient | -0.263 | -0.109
Statistical Analysis 1: Comparison: Alpha Transcranial Alternating Current Stimulation (tACS); Test type: Superiority; p = 0.464, Pearson's correlation
Statistical Analysis 2: Comparison: Sham Stimulation; Test type: Superiority; p = 0.765, Pearson's correlation

4. Secondary Outcome: Correlation Between Changes in the Amplitude of Left Frontal Alpha Oscillations From Baseline to Two-week Follow-up and Depression Symptoms.
Description: Correlation Coefficient (r) will be used to determine if there is a relationship between the change in Hamilton Depression Rating Scale (HDRS) scores from baseline, Day 5 and to two-week follow up and change in the amplitude of left frontal alpha oscillations before stimulation at baseline and Day 5 of stimulation. The HDRS is a clinician-rated measure of depression severity where higher scores indicate greater depression severity. To calculate the amplitude of left frontal alpha oscillations, Fourier transform is applied to 2 second epochs of resting-state EEG data and averaged across epochs. The amplitude of alpha oscillations is calculated and averaged across left frontal electrodes.
Time Frame: Baseline, two-week follow-up visit
Population: Data for 1 participant unavailable due to missed visit.
Measure: Number; unit: Pearson Correlation Coefficient
Arm/Group | Alpha Transcranial Alternating Current Stimulation (tACS) | Sham Stimulation
Number analyzed (Participants) | 9 | 10
Pearson Correlation Coefficient | 0.624 | 0.087
Statistical Analysis 1: Comparison: Alpha Transcranial Alternating Current Stimulation (tACS); Test type: Superiority; p = 0.072, Pearson's correlation
Statistical Analysis 2: Comparison: Sham Stimulation; Test type: Superiority; p = 0.811, Pearson's correlation

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed at Day 1, Day 2, Day 3, Day 4, Day 5 and 2-week follow-up
Arm/Group | Alpha Transcranial Alternating Current Stimulation (tACS) | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alpha Transcranial Alternating Current Stimulation (tACS) (N=10) | Sham Stimulation (N=10)
Headache (Nervous system disorders) | 7 (14) | 7 (27)
Restlessness (Nervous system disorders) | 6 (13) | 3 (6)
Vision Changes (Nervous system disorders) | 1 (1) | 3 (4)
Pain (Musculoskeletal and connective tissue disorders) | 2 (8) | 2 (6)
Nausea (Nervous system disorders) | 0 (0) | 5 (7)
Fatigue (Nervous system disorders) | 7 (25) | 9 (28)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1) | 2 (5)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Eye Twitching (Eye disorders) | 1 (1) | 0 (0)
Vivid Dreams (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT03994081/Prot_SAP_000.pdf